CLINICAL TRIAL: NCT04504708
Title: A Phase 1/2a, Dose-Escalation and Dose-Expansion Study of ZX-101A in Patients With Relapsed/Resistant or Refractory Advanced Hematologic Malignancies
Brief Title: Dose-Escalation and Dose-Expansion Study of ZX-101A in Patients With Relapsed/Resistant or Refractory Advanced Hematologic Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to business decision.
Sponsor: Hangzhou Zenshine Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZX-101A-101
Record Dates: First submitted 2020-07-25; First posted 2020-08-07 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Non-hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ZX-101A Dose Level 1 (Experimental): Starting dose (SD) of ZX-101A administered orally once daily in a 28-day cycle
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level 2 (Experimental): 2-times the SD of ZX-101A administered orally once daily in a 28-day cycle
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level 3 (Experimental): 3-times the SD of ZX-101A administered orally once daily in a 28-day cycle
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level 4 (Experimental): 4-times the SD of ZX-101A administered orally once daily in a 28-day cycle
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level 5 (Experimental): 5-times the SD of ZX-101A administered orally once daily in a 28-day cycle
  Interventions: Drug: ZX-101A

INTERVENTIONS:
Drug: ZX-101A — Once daily, oral dosing of ZX-101A at the assigned dose level for 28 consecutive days in a 28-day cycle

SUMMARY:
ZX-101A-101 is a Phase 1/2a, first-in-human, open-label, multicenter, multiple-ascending dose study to investigate the safety, tolerability, pharmacokinetics, pharmacodynamic, and preliminary antitumor activity of ZX-101A administered orally (PO) once daily (QD) in 28-day cycles in patients with relapsed/resistant or refractory advanced hematologic malignancies [Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL), indolent NHL, and other NHL subtypes).

DETAILED DESCRIPTION:
The ZX-101A-101 study will consist of 2 parts:

* Part 1: ZX-101A Dose Escalation
* Part 2: ZX-101A Dose Expansion

The Part 1 (dose escalation) of the study is designed to determine the safety and tolerability of ZX-101A administered orally once daily in 28-day cycles. The Part 2 (dose expansion) of the study is designed to further investigate the safety, tolerability, pharmacokinetics and pharmacodynamic and clinical activities of ZX-101A administered orally once daily in 28-day cycles at the selected recommended Phase 2 dose (RP2D).

Results of clinical findings in patients in the dose-escalation portion of the study will be reviewed to identify conditions (or genetic characteristics) most likely to respond to ZX-101A. These select types of hematologic malignancies will be enrolled in cohorts in the dose-expansion part of the study.

Male or female patients who are 18 years of age or older with relapsed/resistant or refractory advanced hematologic malignancies (CLL/SLL, iNHL, and other NHL subtypes) will be included in the study provided that all inclusion and exclusion criteria are satisfied.

Up to three cohorts are planned in Part 2 - Dose Expansion of the study: 1) relapsed/resistant or refractory Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL), 2) relapsed/resistant or refractory indolent Non- Hodgkin's Lymphoma (iNHL), and based on emerging data from Part 1-Dose Expansion, a third cohort consisting of other types of NHL may be included.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are ≥ 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Failed at least 2 prior systemic standard therapies.
* Histopathological confirmed diagnosis of CLL/SLL, indolent NHL,and other NHL subtypes.
* Documented active disease that is relapsed/resistant or refractory requiring treatment after established therapy shown to have clinical benefit.
* Acceptable bone marrow, kidney, and liver function.
* No transfusion or cytokine support for ≥ 2 weeks before initiating study treatment.
* Ability to swallow and retain oral medications (see exclusion criteria #20 below).
* Negative serum pregnancy test in women of childbearing potential at Screening.
* Women of childbearing potential and men who partner with a woman of childbearing potential must agree to use effective contraceptive methods.
* Men must agree to no sperm donations during the study and for 3 months after the last dose of ZX-101A.
* Understands the requirements of the study (e.g. periodic imaging studies, periodic blood sampling, bone marrow studies), is willing to comply with all study procedures and signed the Institutional Review Board (IRB)-approved informed consent.

Exclusion Criteria:

* Received investigational study drug within 28 days (or 5 half-lives, whichever is longer).
* Concurrent participation in another therapeutic treatment trial.
* Received approved anti-cancer drugs within 21 days (42 days for nitrosoureas) or 5 half-lives, whichever is longer.
* Ongoing immunosuppression for chronic conditions.
* Known active hepatitis B virus (HBV), hepatitis C virus (HCV), or HIV infection.
* Any concurrent uncontrolled illness.
* Has not recovered from adverse events from prior anti-cancer treatment (with exception of alopecia).
* Pregnant or breast-feeding or planning to conceive or father children within the projected duration of the study.
* Major surgery within 4 weeks prior to first dose of study treatment.
* Radiation treatment within 2 weeks prior to first dose of study treatment.
* Gastrointestinal dysfunction, including motility or malabsorption syndromes or inflammatory bowel disease which could limit absorption of study drug.
* Active or prior pneumonitis or interstitial lung disease.

Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Defining the recommended Phase 2 dose (RP2D) of ZX-101A. | From Day 1 of Cycle 1 through the end of the DLT evaluation period (28 days for the first two Dose Levels and 84 days for Dose Levels 3, 4 and 5); each cycle is 28 days.
  To assess number of patients experiencing dose-limiting toxicities (DLTs) in Part 1.
Safety and tolerability of ZX-101A | From first dose of ZX-101A through 28 days after the last ZX-101A treatment (up to 2 years); each cycle is 28 days.
  To examine the incidence of clinical and laboratory adverse events after multiple doses of ZX-101A in Parts 1 and 2

SECONDARY OUTCOMES:
Peak Plasma Concentration of ZX-101A | Days 1, 2, 15 and 16 of Cycle 1 (each cycle is 28 days), and Day 1 of Cycle 3 and Cycle 5
  To evaluate the maximum observed concentration (Cmax) after single and repeated oral, once daily doses of ZX-101A
Area under the plasma concentration of ZX-101A | Days 1, 2, 15 and 16 of Cycle 1 (each cycle is 28 days), and Day 1 of Cycle 3 and Cycle 5
  To evaluate the area under the curve (AUC) plasma-concentration after single and repeated oral, once daily doses of ZX-101A
Half-life of ZX-101A | Days 1, 2, 15 and 16 of Cycle 1 (each cycle is 28 days), and Day 1 of Cycle 3 and Cycle 5
  To evaluate the half-life of ZX-101A after single and repeated oral, once daily doses of ZX-101A
Phospho-AKT (p-AKT) levels in whole blood | Days 1 and 2 of Cycle 1 (each cycle is 28 days)
  To evaluate the differences phospho-AKT (p-AKT) levels in whole blood before and after single oral dose of ZX-101A.
Objective response rate (ORR) | Up to 2 years
  To evaluate the objective response rate (ORR) as determined by the specific disease response criteria
Duration of response (DoR) | Up to 2 years
  To examine the duration of response (DoR), defined as time from the date of first documentation of response to the date of the first documentation of progressive disease (PD), or death due to any cause
Progression free survival (PFS) | Up to 2 years
  To examine the the progression free survival (PFS), defined as time from the date of first dose of study treatment to the first date of documentation of PD, or death due to any cause
Overall survival (OS) | Up to 2 years
  To examine the overall survival (OS), defined as time from the date of first dose of study treatment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Qin, PhD, Study Director — Zenshine Pharmaceutical, Inc.
Locations (6):
- United States (6):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - ACRC/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Innovative Clinical Research Institute, Long Beach, California
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - University of Toledo Precision Oncology Research, Toledo, Ohio
  - Seattle Cancer Care Alliance, Seattle, Washington